CLINICAL TRIAL: NCT06486753
Title: Effect of Lateral Soft Tissue Release on Patient-Reported Outcomes and Hallux Valgus Angle Correction in Chevron Osteotomy
Brief Title: LSTR in Chevron Osteotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Kevin Varner, Chairman of the Department of Orthopedics, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00026261
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Bunion
MeSH Terms: conditions — Bunion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chevron osteotomy bunion surgery without LSTR (No Intervention): Participants randomized to this group will receive a standard Chevron osteotomy bunion surgery.
- Chevron osteotomy bunion surgery with LSTR (Experimental): Participants randomized to this group will receive a Chevron osteotomy bunion surgery and a lateral soft tissue release.
  Interventions: Procedure: Chevron osteotomy bunion surgery with lateral soft tissue release

INTERVENTIONS:
Procedure: Chevron osteotomy bunion surgery with lateral soft tissue release — Lateral soft tissue release is often performed in hallux valgus correction, and there is preliminary evidence to suggest it may be useful in improving post-surgical outcomes for the Chevron osteotomy bunion surgery.
  Arms: Chevron osteotomy bunion surgery with LSTR

SUMMARY:
The goal of this clinical trial is to determine if performing a lateral soft tissue release during a Chevron osteotomy (or Akin osteotomy when appropriate) for bunions leads to better correction without added complications in 200 patients over the age of 18 years old with the capacity to consent and mild to moderate bunions that are determined to benefit from Chevron osteotomies by one of the IRB approved study physicians. The main questions it aims to answer are:

How does the addition of a lateral soft tissue release (LSTR) in a Chevron osteotomy bunion surgery affect hallux valgus alpha angle (HVA) correction? How does the addition of an LSTR in a Chevron osteotomy bunion surgery affect intermetatarsal angle (IMA) degrees of correction? Researchers will compare Chevron osteotomy bunion surgeries with and without LSTR to see if LSTRs lead to better correction without added complications.

Participants will:

* Be randomized to a control group where they receive a typical Chevron osteotomy bunion surgery or to the experimental group where they receive a Chevron osteotomy bunion surgery with an LSTR.
* Complete surveys preoperatively and at 3, 6, and 12 months after surgery.
* Receive routine x-rays pre and postoperatively to compare hallux valgus angle (HVA).

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years old
* Have mild to moderate bunions that are determined to benefit from Chevron osteotomies

Exclusion Criteria:

* Under the age of 18
* Connective tissue disease
* Juvenile bunions
* Severe bunions
* Revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
Hallux valgus alpha angle correction | Pre-surgery, 6 weeks post surgery

SECONDARY OUTCOMES:
Intermetasarsal angle (IMA) degrees of correction | 3 months, 6 months, and 12 months post surgery
Recurrence of hallux valgus deformity | 3 months, 6 months, and 12 months post surgery
Complications following surgery | 3 months, 6 months, and 12 months post surgery
  We will be looking at complications including possible metatarsal head avascular necrosis (AVN) and over correction (hallux varus).

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States